CLINICAL TRIAL: NCT05296148
Title: A European Feasibility Study of the CroíValve DUO Transcatheter Tricuspid Coaptation Valve System in Patients With Tricuspid Regurgitation
Brief Title: A Feasibility Study of the CroíValve DUO System for Tricuspid Regurgitation
Acronym: TANDEM I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CroiValve Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV005
Record Dates: First submitted 2022-03-07; First posted 2022-03-25 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Treatment with the CroíValve DUO Coaptation Valve System
  Interventions: Device: Transcatheter Tricuspid Valve Implantation

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Implantation — Implantation of a tricuspid coaptation valve through a transcatheter approach.

SUMMARY:
This study is prospective, multicentre, non-randomized single-arm early feasibility study to evaluate the safety and performance of the CroíValve DUO Transcatheter Tricuspid Coaptation Valve System in patients with severe Tricuspid Regurgitation.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of severe Tricuspid Regurgitation per American Society of Echocardiography (ASE) Criteria determined by Echo Core Lab assessment of a qualifying Transthoracic Echocardiogram (TTE).
2. Subject is symptomatic despite medical therapy (NYHA Functional Class II or higher)
3. Subject is on stable medical therapy as assessed by the Heart Team
4. The patient's anatomy is suitable in the judgment of the Investigational Site Heart Team and the Patient Screening Committee.
5. Age ≥18 years
6. The patient or the legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent on a form, as approved by the EC of the respective clinical site.

Exclusion Criteria:

1. Subject is currently participating in another clinical investigation that could affect the outcome of this trial
2. Transesophageal echocardiography (TEE) is contraindicated or unsuccessful
3. Previous tricuspid valve repair, replacement or transcatheter tricuspid intervention
4. Moderate to severe tricuspid valve stenosis
5. Severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation
6. Significant comorbid factors which places the subject at prohibitive risk for surgical repair in the judgment of the Investigational Site Heart Team and the Patient Screening Committee
7. Need for concomitant surgical or interventional procedure known at time of screening (e.g., CABG, Atrial Septal Defect (ASD) repair).
8. Ejection Fraction (EF) <30% within 45 days of the implant procedure
9. Echocardiographic or CT evidence of intracardiac mass, thrombus or vegetation
10. Patient has Systolic Pulmonary Pressure (sPAP) >60 mm Hg
11. Severe hemodynamic instability: cardiogenic shock or the need for inotropic support or Intra-Aortic Balloon Pump (IABP) or other percutaneous ventricular assist devices
12. Severe respiratory instability: Severe COPD or continuous use of home oxygen or has FEV1 <50% of predicted
13. Severe right ventricular dysfunction as determined by the Echo Core Lab
14. Untreated clinically significant coronary artery disease requiring revascularization surgical or interventional PCI
15. Stroke or transient ischemic event within 90 days prior to the implant procedure
16. Untreated severe symptomatic carotid stenosis (>70% by ultrasound)
17. Acute myocardial infarction within 30 days before the index procedure
18. Renal insufficiency (eGFR<25 ml/min)
19. Active endocarditis within 6 months of the implant procedure
20. Pulmonary embolism within the last 6 months
21. Any surgical, interventional, or transcatheter procedure within 30 days prior to the index procedure
22. Patient has an SVC dimension/anatomy is not suitable for device implantation (i.e., extremely tortuous, heavily calcified, aneurysmal)
23. Hypertrophic cardiomyopathy, restrictive cardiomyopathy or constrictive pericarditis
24. Life expectancy <1 year
25. Active infections requiring current antibiotic therapy
26. Known severe liver disease
27. Prior heart or lung transplant
28. Known active peptic ulcer or active GI bleed
29. Unable to take anticoagulant therapy
30. Known patient is actively abusing drugs
31. Subjects who are pregnant or planning to become pregnant
32. Any condition making it unlikely the subject will be able to complete all protocol procedures (including compliance with guideline-directed medical therapy and immobility that would prevent completion of 6MWT), follow-up visits, or impact the scientific soundness of the clinical investigation result
33. Any known major coagulation abnormalities, thrombocytopenia, platelets <50,0000/ml or anemia Hb <9g/dl
34. Any known sensitivities or allergies to contrast and/or the device materials, including nickel and titanium
35. BMI >50kg/m2
36. Transvalvular implanted pacemaker or ICD lead is present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from device or procedure related serious adverse events | Day 30
  Freedom from device or procedure related serious adverse events

SECONDARY OUTCOMES:
Change in TR Grade | Day 30, Month 6, Month 12
  Number of patients with reduction in TR from baseline as assessed by echocardiography
NHYA Functional Class | Day 30, Month 6, Month 12
  Number of patients with improvement in NYHA class
Six Minute Walk Test (6MWT) | Day 30, Month 6, Month 12
  Change in distance (m) from baseline

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne GUMed, Gdansk
  - Górnośląskie Centrum Medyczne im. Prof. Leszka Gieca, Katowice
  - Narodowy Instytut Kardiologii im. Stefana kardynała Wyszyńskiego, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided